CLINICAL TRIAL: NCT04963322
Title: The Incidence and Risk Factors of Biliary Complications in Patients With Extracorporeal Membrane Oxygenation: a Retrospective Observational Study
Brief Title: The Incidence and Risk Factors of Biliary Complications in Patients With ECMO
Status: Completed | Type: Observational
Sponsor: Kim Hee Young (Other)
Responsible Party: Sponsor-Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Organization: Pusan National University Yangsan Hospital (Other)
Other Study IDs: 05-2021-095
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Patients With Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: extracorporeal membrane oxygenation therapy — Extracorporeal membrane oxygenation for the management of severe refractory heart and lung dysfunction

SUMMARY:
By confirming the incidence of biliary tract complications in adult patients aged 18 years or older who received extracorporeal membrane oxygenation , and measuring the duration of application of extracorporeal membrane oxygenation, drugs administered during the application period of extracorporeal membrane oxygenation, duration of fasting period, duration of total intravenous nutrition, and plasma bilirubin concentration, the researchers will try to find risk factors of biliary tract complications in patients receiving extracorporeal membrane oxygenation. Clinically, the researchers will check whether there are modifiable risk factors in patients receiving extracorporeal membrane oxygenation.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation is an important method for the management of severe refractory heart and lung dysfunction, and improvements in extracorporeal membrane oxygenation equipment and increased experience have made it possible to use it for a long time. However, complications following extracorporeal membrane oxygenation are very common, and mortality and morbidity are high. When extracorporeal membrane oxygenation is applied, gastrointestinal bleeding may occur due to stress, ischemia, or bleeding tendency, and direct secondary bilirubin elevation and gallstone formation may occur secondary to long-term fasting, total intravenous nutrition, hemolysis, and diuretics. In intensive care patients, acalculous cholecystitis can progress with multiple organ failure and is known to be associated with prolonged ICU stay and high mortality. However, there is no report on whether the incidence of cholecystitis, risk factors, direct elevation of bilirubin, and cholelithiasis in patients receiving extracorporeal membrane oxygenation progresses to symptomatic cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 who have received extracorporeal membrane oxygenation therapy

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18 who have received extracorporeal membrane oxygenation therapy
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
incidence of biliary tract complications | during application of ECMO (up to 30 days which is the longest duration for applied ECMO)
  incidence of biliary tract complications

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea